CLINICAL TRIAL: NCT03712540
Title: A Drug-Drug Interaction Study to Assess the Effect of Rifampin on the Pharmacokinetics of an Oral Dose of BMS-986278 in Healthy Participants
Brief Title: An Investigational Study of Experimental Medication BMS-986278 Given With the Antibiotic Rifampin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM027-017
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMS-986278 + Rifampin (Experimental): Treatment period A: BMS-986278 alone Treatment period B: Rifampin followed by BMS-986278
  Interventions: Drug: BMS-986278; Drug: Rifampin

INTERVENTIONS:
Drug: BMS-986278 — Oral administration 30 mg
Drug: Rifampin — Oral administration 600 mg

SUMMARY:
The purpose of this study is to investigate the effects of experimental medication BMS-986278 given with the antibiotic Rifampin in healthy participants.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 30.0 kg/m2, inclusive, at screening

Exclusion Criteria:

* Women who are of childbearing potential or breastfeeding
* Any significant acute or chronic medical condition that presents a potential risk to the participant and/or that may compromise the objectives of the study, including active, or history of, liver disease, or intestinal disorder including irritable bowel syndrome
* History or presence of malignancy including hematological malignancies; participants with a history of basal cell or squamous cell carcinoma that has been treated with no evidence of recurrence within 5 years will be allowed for inclusion, as judged by the investigator
* History of significant cardiovascular disease
* Current or recent (within 3 months of study treatment administration) gastrointestinal disease that could impact upon the absorption of study treatment

Other protocol defined inclusion/exclusion criteria could apply

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) for BMS-986278 | Day 1 and 8
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] for BMS-986278 | Up to 24 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] for BMS-986278 | Day 1 and 8
Terminal phase half-life (T-HALF) for BMS-986278 | Day 1 and 8

SECONDARY OUTCOMES:
Incidence of non-serious adverse events (AE) | Up to 24 days
Incidence of serious adverse events (SAE) | Up to 24 days
Incidence of AE leading to discontinuation | Up to 24 days
Incidence of clinically significant changes in vital signs, electrocardiograms (ECGs), physical examinations, and clinical laboratory tests | Up to 24 days
Maximum observed plasma concentration (Cmax) for Rifampin | Day 8
Time of maximum observed plasma concentration (Tmax) for Rifampin | Day 8
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] for Rifampin | Day 8-9
Area under the plasma concentration-time curve from time zero extrapolated to infinite time [AUC(INF)] for Rifampin | Day 8-9

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PRA Health Science KK, Lenexa, Kansas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm